CLINICAL TRIAL: NCT00337090
Title: A Randomized, Double-blind, Parallel Group, Placebo and Active Controlled, Multicenter Dose Ranging Study With the Beta-3 Agonist YM178 in Patients With Symptomatic Overactive Bladder
Brief Title: A Study of YM178 in Patients With Symptomatic Overactive Bladder (DRAGON)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-CL-044
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Overactive Bladder
Keywords: Over Active Bladder; Urinary incontinence; YM178; Symptomatic Over Active Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

INTERVENTIONS:
Drug: YM178

SUMMARY:
The study will examine which dose of YM178 is best in terms of efficacy, safety and tolerability compared to placebo and compared to tolterodine, a marketed product.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years suffering from overactive bladder (OAB) for more than 3 months

Exclusion Criteria:

* Pregnant and breastfeeding women
* Any medical condition or need for co-medication which interferes with the drug under investigation (YM178) or the comparator (tolterodine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1108 (Actual)
Dates: Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma, Study Chair — Astellas Pharma Europe B.V.
Locations (84):
- Belgium (5):
  - 3 Sites, Antwerp
  - 2 Sites, Brussels
  - Ghent
  - Leuven
  - Liège
- Czechia (6):
  - Brno
  - Mělník
  - Ostrava
  - 3 Sites, Prague
  - Ústí nad Labem
  - Zlín
- Denmark (3):
  - Holbæk
  - Kolding
  - Roskilde
- France (2):
  - 2 Sites, Nantes
  - 2 Sites, Paris
- Germany (15):
  - Bad Ems
  - Bamberg
  - Bautzen
  - Berlin
  - Dresden
  - Frankfurt
  - Hagenow
  - Halle
  - Hamburg
  - Koblenz
  - Leipzig
  - München
  - Radebeul
  - Trier
  - Uetersen
- Greece (2):
  - 3 Sites, Athens
  - Pátrai
- Hungary (6):
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Sopron
  - Szeged
  - Tatabánya
- Italy (9):
  - Catanzaro
  - Milan
  - Modena
  - Padua
  - Roma
  - Sassari
  - Torino
  - Udine
  - Varese
- Netherlands (6):
  - Amsterdam
  - Apeldoorn
  - Arnhem
  - Eindhoven
  - Enschede
  - Maastricht
- Norway (3):
  - Bergen
  - Oslo
  - Tønsberg
- Poland (6):
  - Bialystok
  - Katowice
  - Kielce
  - Lublin
  - 3 Sites, Warsaw
  - 3 Sites, Wroclaw
- Russia (2):
  - 7 Sites, Moscow
  - 3 Sites, Saint Petersburg
- Spain (8):
  - 2 Sites, Barcelona
  - Bilbao
  - 2 Sites, Madrid
  - Manacor
  - Miranda de Ebro
  - San Juan de Alica
  - Seville
  - Vigo
- Sweden (2):
  - Gothenburg
  - 2 Sites, Stockholm
- United Kingdom (9):
  - Birmingham
  - Blackburn
  - Chichester
  - Croydon
  - London
  - Reading
  - Sheffield
  - Southampton
  - Swansea

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401